CLINICAL TRIAL: NCT02572219
Title: Effects of a Nutraceutical Preparation on Cognitive Impairment in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Giuseppe Lembo, prof. Giuseppe Lembo, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LMB04
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Nutraceutical (Active Comparator): Treated with nutraceutical compound
  Interventions: Dietary Supplement: Nutraceutical compound
- Placebo (Placebo Comparator): Treated with placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutraceutical compound
  Arms: Nutraceutical
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Aim of this randomized, double-blind clinical study is to evaluate the efficacy of a nutraceutical preparation on early markers of cognitive impairment, in patients affected by arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Males or females between 40 and 65 years of age;
* Hypertensive patients classified according to their SBP (Systolic Blood Pressure) and DBP (Diastolic Blood Pressure) values. Included patients will be those with stage 1 hypertension (SBP 140-159 mmHg; DBP 90-99 mmHg) and with stage 2 hypertension (SBP 160-179 mmHg; DBP 100-109 mmHg).

Exclusion Criteria:

* Previous acute myocardial infarction (AMI);
* Previous stroke and/or transient ischemic attack (TIA);
* Diabetes mellitus;
* History of atrial fibrillation or other severe arrhythmias;
* Severe cardiovascular diseases;
* Renal pathologies (creatinine > 1.4 mg/dL);
* Preexisting psychiatric pathologies;
* Neurodegenerative diseases, such as multiple sclerosis, lateral amyotrophic sclerosis, Parkinson, Alzheimer, neuromuscular pathologies, epilepsy;
* Diagnosis of dementia;
* Depression;
* Long-term regular use of anxiolytics drugs, antidepressant drugs, antipsychotic drugs, hypnoinducing drugs, cognitive stimulators.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Cognitive function assessed by neuropsychological tests | 6 months
  Patients will be subjected to Montreal Cognitive Assessment (MoCA), Verbal fluency test, Word coupling test, Stroop test, and Instrumental Activities of Daily Living - IADL test. Assessments of cognitive functions will be performed by using unique score measurements defined in Units on a Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, (is), Italy